CLINICAL TRIAL: NCT01232023
Title: Evaluation of Pharmacokinetic and Pharmacodynamic Characteristics of Indobufen, an Anticoagulant Agent
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Asan Medical Center, Clinical Pharmacology & Therapeutics, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-0103
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Indobufen; healthy volunteers
MeSH Terms: interventions — indobufen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100mg (Experimental): Wild type UGT1A : 3 / Variant type UGT1A : 3
  Interventions: Drug: Indobufen
- 200mg (Experimental): Wild type UGT1A : 3 / Variant type UGT1A : 3
  Interventions: Drug: Indobufen
- 400mg (Experimental): Wild type UGT1A : 3 / Variant type UGT1A : 3
  Interventions: Drug: Indobufen
- 800mg (Experimental): Wild type UGT1A : 3 / Variant type UGT1A : 3
  Interventions: Drug: Indobufen

INTERVENTIONS:
Drug: Indobufen — Single Oral Dose of

SUMMARY:
This study is designed to evaluate the pharmacokinetic and pharmacodynamic characteristics of indobufen in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 19 to 50 years at screening.
* Subjects with body weight ≥ 45 kg and within ±20% of the ideal body weight : Ideal body weight = (height [cm] - 100)x0.9.
* Subjects who have received and understood completely the information regarding the current study and given written informed consents to voluntarily participate in the study and followed all instructions specified in the protocol.

Exclusion Criteria:

* Subjects who have drunken habitually (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the study period from 2 days prior to the first administration of investigational product and during this study.
* Subjects deemed ineligible by investigator based on other reasons, including abnormal laboratory values or diseases.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics | 24 Hours
  AUC, Cmax

SECONDARY OUTCOMES:
Pharmacodynamics | 24 Hours
  Platelet Aggregation Test

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr